CLINICAL TRIAL: NCT00594074
Title: Alcohol in the Treatment of Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00008809; 7638 (Other: DUMC)
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Obesity, Weight Loss, Alcohol Drinking
MeSH Terms: conditions — Obesity; Weight Loss; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This group will receive 3.25 ounces of white wine with lunch and dinner
  Interventions: Other: white wine
- 2 (No Intervention): This group receives the same amount of calories as the experimental group

INTERVENTIONS:
Other: white wine — 3.25 ounces of white wine twice a day with lunch and dinner
  Arms: 1

SUMMARY:
This pilot study looks at the relationship of moderate alcohol consumption on weight loss.

DETAILED DESCRIPTION:
We hypothesize that individuals who consume a moderate amount of alcohol, such as a glass or two of wine daily, will lose more during a weight-reduction program than will those who do not, if equal calories are administered to both groups. The purpose of this pilot study is to look at the relationship of alcohol in weight loss. The current standard in weight loss programs is to eliminate alcohol from the diet. We propose to enroll 50 females enrolled at the Structure House residential diet program in Durham, North Carolina. Half or the subjects will receive 150 calories in the form of white wine, 3.5 ounce with lunch and 3.5 ounces with dinner. The other half of the subjects wil receive their 150 calories in their regular diet. All participants are asked not to consume any additional alcohol. Participants will be weighed daily. The study lasts four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >21, female, BMI ≥ 30, no history of substance abuse, prior alcohol use of at least one drink/week; Exclusion:
* pregnancy, breast feeding, previous history of alcohol abuse, liver disease.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
An outcome measure for the study is an increase weight loss or no change in the wine group of .05% over the 4 weeks of the study | 4 weeks

SECONDARY OUTCOMES:
Participants will also be asked to complete a visual satiety scale each day before and after lunch and dinner. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Surwit, Ph.D., ABPP,, Principal Investigator — Duke University
Locations (1):
- Structure House, LLC, Durham, North Carolina, United States

REFERENCES:
- [Background] Ajani, U. A., Hennekens, C. H., Spelsberg, A., & Manson, J. E. (2000). Alcohol consumption and risk of type 2 diabetes mellitus among US male physicians. Arch Intern Med, 160(7), 1025-1030. Dallongeville, J., Marecaux, N., Ducimetiere, P., Ferrieres, J., Arveiler, D., Bingham, A., et al. (1998). Influence of alcohol consumption and various beverages on waist girth and waist-to-hip ratio in a sample of French men and women. Int J Obes Relat Metab Disord, 22(12), 1178-1183. Flechtner-Mors, M., Biesalski, H. K., Jenkinson, C. P., Adler, G., & Ditschuneit, H. H. (2004). Effects of moderate consumption of white wine on weight loss in overweight and obese subjects. Int J Obes Relat Metab Disord, 28(11), 1420-1426. Melanson, K. & Dwyer, J. (2002). Popular diets for treatment of overweight and obesity. In T. A. S. Wadden, A. J. (Ed.), Handbook of obesity treatment (2 ed., pp. 249-282). New York: The Guilford Press. Rimm, E. B., Chan, J., Stampfer, M. J., Colditz, G. A., & Willett, W. C. (1995). Prospective study of cigarette smoking, alcohol use, and the risk of diabetes in men. Bmj, 310(6979), 555-559. Stampfer, M. J., Colditz, G. A., Willett, W. C., Manson, J. E., Arky, R. A., Hennekens, C. H., et al. (1988). A prospective study of moderate alcohol drinking and risk of diabetes in women. Am J Epidemiol, 128(3), 549-558. Wannamethee, S. G., Camargo, C. A., Jr., Manson, J. E., Willett, W. C., & Rimm, E. B. (2003). Alcohol drinking patterns and risk of type 2 diabetes mellitus among younger women. Arch Intern Med, 163(11), 1329-1336. Wannamethee, S. G., Field, A. E., Colditz, G. A., & Rimm, E. B. (2004). Alcohol intake and 8-year weight gain in women: a prospective study. Obes Res, 12(9), 1386-1396.